CLINICAL TRIAL: NCT02711137
Title: A Phase 1/2, Open-Label, Dose-Escalation/Dose-Expansion, Safety and Tolerability Study of INCB057643 in Subjects With Advanced Malignancies
Brief Title: Open-Label Safety and Tolerability Study of INCB057643 in Subjects With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated due to safety issues.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 57643-101; 2017-002641-29 (EudraCT Number)
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Results first posted 2022-04-28 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors
Keywords: Solid tumor; lymphoma; leukemia; AML; myelodysplastic syndrome (MDS); multiple myeloma; myeloproliferative neoplasm (MPN); MDS/MPN; myelofibrosis (MF); pancreatic cancer; colorectal cancer; non-small cell lung cancer; prostate cancer; breast cancer; ovarian cancer; glioblastoma multiforme (GBM); NUT midline carcinoma; non-Hodgkin lymphoma; diffuse large B-cell lymphoma (DLBCL); double-hit; triple-hit; myc; bromodomain and extra-terminal (BET) inhibitor
MeSH Terms: conditions — Lymphoma; Leukemia; Myelodysplastic Syndromes; Multiple Myeloma; Myeloproliferative Disorders; Primary Myelofibrosis; Pancreatic Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Glioblastoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse | interventions — INCB057643; Gemcitabine; Paclitaxel; rucaparib; abiraterone; ruxolitinib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part1/Treatment Group A : 8mg QD INCB057643 (Experimental): Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the TGA.
  Treatment Group A included solid tumors and lymphoma
  Interventions: Drug: INCB057643
- Part1/Treatment Group A : 12mg QD INCB057643 (Experimental): Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the TGA.
  Treatment Group A included solid tumors and lymphoma
  Interventions: Drug: INCB057643
- Part1/Treatment Group A : 16mg QD INCB057643 (Experimental): Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the TGA.
  Treatment Group A included solid tumors and lymphoma
  Interventions: Drug: INCB057643
- Part1/Treatment Group B : 8mg QD INCB057643 (Experimental): Initial cohort dose of INCB054763 monotherapy at the protocol-specified cohort escalation treatment group B (TGB), based on protocol-specific criteria. Treatment Group B included any acute leukemia, HRMDS, MDS/MPN, or MF
  Interventions: Drug: INCB057643
- Part1/Treatment Group B : 12mg QD INCB057643 (Experimental): Initial cohort dose of INCB054763 monotherapy at the protocol-specified cohort escalation treatment group B (TGB), based on protocol-specific criteria. Treatment Group B included any acute leukemia, HRMDS, MDS/MPN, or MF.
  Interventions: Drug: INCB057643
- Part1/Treatment Group C : 8mg QD INCB057643 (Experimental): Initial cohort dose of INCB054763 monotherapy at the protocol-specified cohort escalation treatment group C (TGC), based on protocol-specific criteria. Treatment Group C includes subjects with MM
  Interventions: Drug: INCB057643
- Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort (Experimental): Initial cohort dose of INCB054763 monotherapy at the specified RP2D dose selected in Part 1 cohort escalation treatment group A (TGA), based on protocol-specific criteria. Part 2 Treatment Group A expansion included pancreatic adenocarcinoma, castration-resistant prostrate cancer, breast cancer, high grade serious ovarian cancer, glioblastoma multiform, non-hodgkin's lymphoma, ewing's sarcoma, and solid tumor or lymphoma.
  Interventions: Drug: INCB057643
- Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort (Experimental): Initial cohort dose of INCB057463 monotherapy at the specified RP2D dose selected in Part 1 cohort escalation treatment group B (TGB), based on protocol-specific criteria. Part 2 Treatment Group B expansion included pancreatic adenocarcinoma, castration-resistant prostrate cancer, breast cancer, high grade serious ovarian cancer, glioblastoma multiform, non-hodgkin's lymphoma, ewing's sarcoma, and solid tumor or lymphoma.
  Interventions: Drug: INCB057643
- Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg (Experimental): Initial cohort dose of INCB057643 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Gemcitabine) in relapsed or refractory advanced or metastatic solid tumors and hematologic malignancies where Gemcitabine is relevant
  Interventions: Drug: INCB057643; Drug: Gemcitabine
- Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg (Experimental): Initial cohort dose of INCB054763 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Paclitaxel) in relapsed or refractory advanced or metastatic solid tumors and hematologic malignancies.
  Interventions: Drug: INCB057643; Drug: Paclitaxel
- Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg (Experimental): Initial cohort dose of INCB054763 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Rucaparib) in relapsed or refractory advanced or metastatic solid tumors and hematologic malignancies.
  Interventions: Drug: INCB057643; Drug: Rucaparib
- Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni (Experimental): Initial cohort dose of INCB054763 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Abiraterone + Prednisone) in Castration Resistant Prostrate Cancer
  Interventions: Drug: INCB057643; Drug: Abiraterone
- Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg (Experimental): Initial cohort dose of INCB054763 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Ruxolitinib) in Myelofibrosis.
  Interventions: Drug: INCB057643; Drug: Ruxolitinib
- Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg (Experimental): Initial cohort dose of INCB054763 monotherapy based on protocol-specific criteria. Part 3 will determine the MTD and/or a tolerated dose of the combination of INCB057643 and one of the SOC agents (Azacitidine) in Acute Myeloid Leukemia and Myelodysplastic Syndrome
  Interventions: Drug: INCB057643; Drug: Azacitidine

INTERVENTIONS:
Drug: INCB057643 — Initial cohort dose of INCB057643 at the protocol-specified starting dose (Part 1), with subsequent dose escalations based on protocol-specific criteria. The recommended treatment group-specific dose(s) will be taken forward into expansion cohorts (Part 2).
Drug: Gemcitabine — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg
Drug: Paclitaxel — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg
Drug: Rucaparib — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg
Drug: Abiraterone — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni
Drug: Ruxolitinib — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg
Drug: Azacitidine — Standard of Care (SOC) agents
  Arms: Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg

SUMMARY:
The purpose of the Study is to select a dose and assess the safety and tolerability of INCB057643 as a monotherapy (Part 1 and Part 2) and in combination with standard-of-care (SOC) agents (Part 3 and Part 4) for subjects with advanced malignancies.

Part 1 will determine the maximum tolerated dose of INCB057643 and/or a tolerated dose that demonstrates sufficient pharmacologic activity. Part 2 will further evaluate the safety, preliminary efficacy, PK, and PD of the dose(s) selected in Part 1 in select tumor types including solid tumors, lymphomas and other hematologic malignancies. Part 3 will determine the tolerated dose of INCB057643 in combination with select SOC agents; and assess the safety and tolerability of the combination therapy in select advanced solid tumors and hematologic malignancies. Part 4 will further evaluate the safety, preliminary efficacy, PK, and PD of the selected dose combination from Part 3 in 4 specific advanced solid tumor and hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of relapsed or refractory advanced or metastatic malignancies:

  * Part 1: solid tumors or lymphomas, or hematologic malignancies
  * Part 2: histologically confirmed disease in specific tumor types
  * Part 3: advanced solid tumor or hematologic malignancy
  * Part 4: select advanced solid tumor or hematologic malignancy
* For Part 1 and 2, subjects must have progressed following at least 1 line of prior therapy and there is no further established therapy that is known to provide clinical benefit (including subjects who are intolerant to the established therapy)
* For Parts 3 and 4, subjects must have progressed following at least 1 line of prior therapy, and the treatment with the select SOC agent is relevant for the specific disease cohort.
* Life expectancy > 12 weeks, for MF subjects in Parts 3 and 4, life expectancy > 24 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status

  * Parts 1 and 3: 0 or 1
  * Parts 2 and 4: 0, 1, or 2
* Willingness to avoid pregnancy or fathering children

Exclusion Criteria:

* Inadequate bone marrow function per protocol-specified hemoglobin, platelet count, and absolute neutrophil count
* Inadequate organ function per protocol-specified total bilirubin, AST and ALT, creatinine clearance and alkaline phosphatase.
* Receipt of anticancer medications or investigational drugs within protocol-specified intervals
* Unless approved by the medical monitor, may not have received an allogeneic hematopoietic stem cell transplant within 6 months before treatment, or have active graft-versus-host-disease following allogeneic transplant
* Unless approved by the medical monitor, may not have received autologous hematopoietic stem cell transplant within 3 months before treatment
* Any unresolved toxicity ≥ Grade 2 (except stable Grade 2 peripheral neuropathy or alopecia) from previous anticancer therapy
* Radiotherapy within the 2 weeks before initiation of treatment. Palliative radiation treatment to nonindex or bone lesions performed less than 2 weeks before treatment initiation may be considered with medical monitor approval
* Currently active and uncontrolled infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment
* Untreated brain or central nervous system (CNS) metastases or brain/CNS metastases that have progressed
* History or presence of abnormal electrocardiogram (ECG) that, in the investigator's opinion, is clinically meaningful
* Type 1 diabetes or uncontrolled Type 2 diabetes
* HbA1c of ≥ 8% (all subjects will have HbA1c test at screening)
* Any sign of clinically significant bleeding
* Coagulation panel within protocol-specified parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, PhD, Study Director — Incyte Corporation
Locations (18):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - University of California, La Jolla, California
  - Sarah Cannon Research Institute at Health One, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Hematology - Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - University of Rochester, Wilmot Cancer Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oncology Consultants, P.A., Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Institut Jules Bordet, Clinical Trial Conduct Unit, Brussels, Belgium
- HÔPITAL SAINT-LOUIS, Service Hématologie Adultes, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchook G, Rosen S, LoRusso P, Watts J, Gupta S, Coombs CC, Talpaz M, Kurzrock R, Mita M, Cassaday R, Harb W, Peguero J, Smith DC, Piha-Paul SA, Szmulewitz R, Noel MS, Yeleswaram S, Liu P, Switzky J, Zhou G, Zheng F, Mehta A. Development of 2 Bromodomain and Extraterminal Inhibitors With Distinct Pharmacokinetic and Pharmacodynamic Profiles for the Treatment of Advanced Malignancies. Clin Cancer Res. 2020 Mar 15;26(6):1247-1257. doi: 10.1158/1078-0432.CCR-18-4071. Epub 2019 Sep 16. PMID 31527168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 137 subjects enrolled at 19 different sites in USA.
Pre-assignment Details: Subjects were assigned to either dose escalation/dose-expansion study of INCB057643 as monotherapy or in combination with SOC agents in subjects with relapsing or refractory malignancies.
Groups:
- Enrolled But Not Dosed: 3 participants enrolled in the study and discontinued the study before study drug is administered
Period: Overall Study
Arm/Group | Part1/Treatment Group A : 8mg QD INCB057643 | Part1/Treatment Group A : 12mg QD INCB057643 | Part1/Treatment Group A : 16mg QD INCB057643 | Part1/Treatment Group B : 8mg QD INCB057643 | Part1/Treatment Group B : 12mg QD INCB057643 | Part1/Treatment Group C : 8mg QD INCB057643 | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg | Enrolled But Not Dosed
Started | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2 | 3
Not completed — Death | 1 | 4 | 5 | 5 | 3 | 1 | 61 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 1 | 1 | 0 | 12 | 2 | 1 | 1 | 3 | 2 | 1 | 1 | 2
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 1 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part1/Treatment Group A : 8mg QD INCB057643 | Part1/Treatment Group A : 12mg QD INCB057643 | Part1/Treatment Group A : 16mg QD INCB057643 | Part1/Treatment Group B : 8mg QD INCB057643 | Part1/Treatment Group B : 12mg QD INCB057643 | Part1/Treatment Group C : 8mg QD INCB057643 | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg | Enrolled But Not Dosed | Total
Number analyzed (Participants) | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2 | 3 | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (10.21) | 60.2 (12.26) | 60.5 (11.44) | 68.9 (5.81) | 75.8 (7.33) | 70.0 (NA) — SD is not calculable as there is only 1 participant enrolled in this arm. | 60.6 (13.80) | 72.6 (10.92) | 72.0 (0) | 56.0 (12.73) | 66.0 (6.16) | 67.7 (4.04) | 75.0 (0) | 76.5 (2.12) | 66.0 (6.24) | 63.0 (12.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 3 | 1 | 0 | 48 | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 1 | 68
  Male | 2 | 3 | 3 | 4 | 4 | 1 | 38 | 5 | 0 | 1 | 0 | 3 | 1 | 2 | 2 | 69
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 3 | 3 | 5 | 6 | 4 | 0 | 71 | 5 | 0 | 1 | 4 | 3 | 1 | 2 | 3 | 111
  Black/African American | 1 | 0 | 2 | 1 | 0 | 0 | 10 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 16
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American-Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian/Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE's).
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Time Frame: From screening through at least 30 days after end of treatment, up to approximately 24 months
Population: All participants enrolled in the study who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part1/Treatment Group A : 8mg QD INCB057643 | Part1/Treatment Group A : 12mg QD INCB057643 | Part1/Treatment Group A : 16mg QD INCB057643 | Part1/Treatment Group B : 8mg QD INCB057643 | Part1/Treatment Group B : 12mg QD INCB057643 | Part1/Treatment Group C : 8mg QD INCB057643 | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg
Number analyzed (Participants) | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2
Participants | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2

2. Secondary Outcome: Percent Inhibition of Total Cellular Myc Protein Concentrations Before and After Administration of INCB057643 When Administered as Monotherapy in an Ex-vivo Assay
Description: An ex vivo assay (utilized in monotherapy only), Measuring Total c-Myc protein expressed from an exogenously added cell line (KMS12BM) to patient plasma, before and after administration of INCB057643.
Time Frame: PD in plasma at pre-dose and 0.5, 1, 2, 4, 6 and 8 hours postdose, for C1D1 and C1D8, and 24hrs post dose for C1D1
Measure: Mean (Standard Error); unit: %Inhibition of Total c-Myc
Groups:
- 8mg QD INCB057643: cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA,TGB,TGC.
- 12mg QD INCB057643: 12mg QD INCB057643 Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA,TGB, and Part 2 TGA,TGB.
- 16mg QD INCB057643: Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA
Arm/Group | 8mg QD INCB057643 | 12mg QD INCB057643 | 16mg QD INCB057643
Number analyzed (Participants) | 11 | 51 | 7
%Inhibition of Total c-Myc
  C1D1 | 24 (199.5) | 28 (200.1) | 54 (236.3)
  C1D8 | 30 (42.59) | 43.4 (52.7) | 65 (55.21)

3. Secondary Outcome: Objective Response Rate (ORR) With INCB057643 in Solid Tumors
Description: Objective response rate is defined as the proportion of subjects who have an objective response using the applicable disease assessment criteria. ORR was proportion of participants with best overall response [complete response (CR) or partial response (PR)].
Time Frame: Efficacy measures from screening through end of treatment and follow-up (every 9 weeks), up to approximately 24 months
Population: The efficacy evaluable population included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Part1/Treatment Group A : 8mg QD INCB057643 | Part1/Treatment Group A : 12mg QD INCB057643 | Part1/Treatment Group A : 16mg QD INCB057643 | Part1/Treatment Group B : 8mg QD INCB057643 | Part1/Treatment Group B : 12mg QD INCB057643 | Part1/Treatment Group C : 8mg QD INCB057643 | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg
Number analyzed (Participants) | 4 | 5 | 8 | 7 | 5 | 1 | 86 | 5 | 1 | 2 | 4 | 3 | 1 | 2
Participants
  Solid Tumors: number analyzed (Participants) | 3 | 4 | 6 | 0 | 0 | 0 | 63 | 0 | 1 | 2 | 4 | 3 | 0 | 0
  Solid Tumors | 0 | 0 | 0 |  |  |  | 0 |  | 0 | 1 | 0 | 0 |  |
  Lymphoma: number analyzed (Participants) | 1 | 1 | 2 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphoma | 1 | 0 | 1 |  |  |  | 2 |  |  |  |  |  |  |
  AML: number analyzed (Participants) | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 2
  AML |  |  |  | 0 | 0 |  |  | 1 |  |  |  |  |  | 0
  Glioblastoma: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Glioblastoma |  |  |  |  |  |  | 0 |  |  |  |  |  |  |
  Myelodysplastic Syndrome: number analyzed (Participants) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Myelodysplastic Syndrome |  |  |  | 0 | 0 |  |  | 0 |  |  |  |  |  |
  Myelofibrosis: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Myelofibrosis |  |  |  | 0 |  |  |  | 0 |  |  |  |  | 0 |
  Multiple Myeloma: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Multiple Myeloma |  |  |  |  |  | 0 |  |  |  |  |  |  |  |

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of INCB057643.
Description: Maximum Observed Plasma Concentration INCB057643 administered as monotherapy in fasted state.
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 hours on C1D1 and C1D8
Population: PK evaluable population includes all subjects who received at least 1 dose of study drug and had at least 1 PK sample collected and analyzed
Measure: Mean (Standard Deviation); unit: nM
Groups:
- 8mg QD INCB057643: Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA,TGB,TGC, and Part 2 TGA
- 12mg QD INCB057643: Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA,TGB, and Part 2 TGA,TGB.
Arm/Group | 8mg QD INCB057643 | 12mg QD INCB057643 | 16mg QD INCB057643
Number analyzed (Participants) | 12 | 99 | 7
nM
  C1D1 | 201 (83.6) | 266 (94.7) | 343 (93.2)
  C1D8: number analyzed (Participants) | 10 | 89 | 7
  C1D8 | 210 (93.2) | 293 (113) | 340 (165)

5. Secondary Outcome: Tmax: Time to Maximum Plasma Concentration of INCB057643
Description: Time to maximum plasma concentration of INCB057643 administered as monotherapy in fasted state
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 hours on C1D1 and C1D8
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Groups:
- 12mg QD INCB057643: Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the Part 1 TGA,TGB, and Part 2 TGA
Arm/Group | 8mg QD INCB057643 | 12mg QD INCB057643 | 16mg QD INCB057643
Number analyzed (Participants) | 12 | 99 | 7
hours
  C1D1 | 2.00 [1.00 to 24.00] | 2 [0.50 to 8.00] | 2.00 [2.00 to 4.00]
  C1D8: number analyzed (Participants) | 10 | 89 | 7
  C1D8 | 1.00 [1.00 to 4.00] | 2 [0.50 to 8.00] | 2.00 [2.00 to 4.00]

6. Secondary Outcome: AUC0-t: Area Under the Single-dose Plasma Concentration-time Curve of INCB057643
Description: Area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration of INCB057643 administered as monotherapy in fasted state
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 hours on C1D1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | 8mg QD INCB057643 | 12mg QD INCB057643 | 16mg QD INCB057643
Number analyzed (Participants) | 12 | 99 | 7
h*nM | 2090 (50.1) | 2550 (39.5) | 3210 (34.3)

7. Secondary Outcome: AUC0-24: Area Under the Steady-state Plasma Concentration-time Curve of INCB057643 Administered as Monotherapy
Description: Area under the steady-state plasma concentration-time curve over 1 dosing interval from Hour 0 to 24 for QD administration of INCB057643 administered as monotherapy in fasted state
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8 hours on C1D8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | 8mg QD INCB057643 | 12mg QD INCB057643 | 16mg QD INCB057643
Number analyzed (Participants) | 10 | 89 | 7
h*nM | 1940 (45.1) | 2740 (43.2) | 3610 (71.9)

8. Secondary Outcome: Part 2 - Cmax: Maximum Observed Plasma Concentration of INCB057643.
Description: Maximum Observed Plasma Concentration INCB057643 administered as monotherapy in fed state.
Time Frame: C2D1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nM
Groups:
- 12mg QD INCB057643: Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in Part 2 TGA and TGB
Arm/Group | 12mg QD INCB057643
Number analyzed (Participants) | 11
nM | 220 (32.0)

9. Secondary Outcome: Part 2-Tmax: Time to Maximum Plasma Concentration of INCB057643
Description: Time to maximum plasma concentration of INCB057643 administered as monotherapy in fed state
Time Frame: C2D1
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | 12mg QD INCB057643
Number analyzed (Participants) | 11
hours | 6.00 [4.00 to 8.00]

10. Secondary Outcome: AUC0-24: Area Under the Steady-state Plasma Concentration-time Curve of INCB057643 Administered as Monotherapy
Description: Area under the steady-state plasma concentration-time curve over 1 dosing interval from Hour 0 to 24 for QD administration of INCB057643 administered as monotherapy in fed state.
Time Frame: C2D1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | 12mg QD INCB057643
Number analyzed (Participants) | 11
h*nM | 2980 (31.5)

ADVERSE EVENTS:
Time Frame: From screening through at least 30 days after end of treatment, up to approximately 24 months
Groups:
- Part1/Treatment Group A : 8mg QD INCB057643: Part1/Treatment Group A : 8mg QD INCB057643 Initial cohort dose of INCB057643 monotherapy at the protocol specified starting dose in the TGA.
  Treatment Group A included solid tumors and lymphoma
Arm/Group | Part1/Treatment Group A : 8mg QD INCB057643 | Part1/Treatment Group A : 12mg QD INCB057643 | Part1/Treatment Group A : 16mg QD INCB057643 | Part1/Treatment Group B : 8mg QD INCB057643 | Part1/Treatment Group B : 12mg QD INCB057643 | Part1/Treatment Group C : 8mg QD INCB057643 | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg
All-Cause Mortality (participants affected / at risk) | 2/4 | 4/5 | 5/8 | 6/7 | 4/5 | 1/1 | 68/86 | 3/5 | 0/1 | 1/2 | 1/4 | 1/3 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/5 | 4/8 | 5/7 | 4/5 | 1/1 | 32/86 | 4/5 | 0/1 | 0/2 | 0/4 | 1/3 | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 7/8 | 7/7 | 5/5 | 0/1 | 82/86 | 5/5 | 1/1 | 2/2 | 4/4 | 3/3 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1/Treatment Group A : 8mg QD INCB057643 (N=4) | Part1/Treatment Group A : 12mg QD INCB057643 (N=5) | Part1/Treatment Group A : 16mg QD INCB057643 (N=8) | Part1/Treatment Group B : 8mg QD INCB057643 (N=7) | Part1/Treatment Group B : 12mg QD INCB057643 (N=5) | Part1/Treatment Group C : 8mg QD INCB057643 (N=1) | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort (N=86) | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort (N=5) | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg (N=1) | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg (N=2) | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg (N=4) | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni (N=3) | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg (N=1) | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus oesophagitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part1/Treatment Group A : 8mg QD INCB057643 (N=4) | Part1/Treatment Group A : 12mg QD INCB057643 (N=5) | Part1/Treatment Group A : 16mg QD INCB057643 (N=8) | Part1/Treatment Group B : 8mg QD INCB057643 (N=7) | Part1/Treatment Group B : 12mg QD INCB057643 (N=5) | Part1/Treatment Group C : 8mg QD INCB057643 (N=1) | Part2/Treatment Group A : 12 mg INCB057643 Expansion Cohort (N=86) | Part2/Treatment Group B : 12 mg INCB057643 Expansion Cohort (N=5) | Part3/Treatment Group A : 8 mg INCB057643 + Gemcitabine 1000mg (N=1) | Part3/Treatment Group B : 8 mg INCB057643 + Paclitaxel 80mg (N=2) | Part3/Treatment Group C : 8 mg INCB057643 + Rucaparib 600mg (N=4) | Part3/Treatment Group D : 8 mg INCB057643 + Abir +Predni (N=3) | Part3/Treatment Group E : 8 mg INCB057643 + Ruxolitinib 20mg (N=1) | Part3/Treatment Group F : 8 mg INCB057643 + Azacitidine 75mg (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 3 (3) | 4 (4) | 3 (9) | 0 (0) | 15 (17) | 4 (11) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chancroid (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 19 (19) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 10 (12) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 27 (28) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 11 (15) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 21 (25) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (12) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 16 (16) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 9 (9) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (9) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 36 (41) | 3 (3) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 13 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 4 (4) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 43 (47) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (6) | 5 (6) | 1 (1) | 0 (0) | 19 (26) | 3 (3) | 0 (0) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 26 (35) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT02711137/Prot_SAP_000.pdf